CLINICAL TRIAL: NCT03071367
Title: Title: A Comparison of Clinical Simulation and Classical Learning for Airway Management in Medical Students: a Randomized Controlled Trial
Brief Title: A Comparison of Clinical Simulation and Classical Learning for Airway Management in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Leopoldo Ferrer, Anesthesiologist, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCEI-1357-2012
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Educational Activities
Keywords: Airway Management; Medical students; Intratracheal intubation; Educational Technology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Simulation (Experimental)
  Interventions: Other: Clinical Simulation
- Classical Learning (No Intervention)

INTERVENTIONS:
Other: Clinical Simulation
  Arms: Clinical Simulation

SUMMARY:
Multiple studies have shown clinical simulation benefits over classical learning method. Research on simulation of airway management has focused on endotracheal intubation training, while research on ventilation via facemask is scant. The investigators compared both learning methods regarding the acquirement of basic skills for airway management by medical students. Students in the clinical simulation group received a 3-hour training on airway management on the first day of their 28-day anesthesia rotation, while classical learning did not. On the last day of rotation, participants were evaluated based on a validated instrument of scores. Primary outcome was airway management scores. Secondary outcomes were rate of success of intubation and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Last year medical students at Universidad de los Andes
* Over 18 year old

Exclusion Criteria:

* Previous elective anesthesia rotation
* Motor deficit affecting the upper limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-06-20 (Actual)

PRIMARY OUTCOMES:
Airway management score | 28 days

SECONDARY OUTCOMES:
Successful intubation rate | 28 days
Incidence of complications | 28 days

IPD SHARING:
Plan to Share IPD: No